CLINICAL TRIAL: NCT01078311
Title: Phase 2 Study of Measurement of Trough Levels of Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Brief Title: Drug Monitoring of Sorafenib in Patients With Advanced Hepatocellular Carcinoma
Acronym: DOSE-HEP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: South West Sydney Local Health District (Other)
Responsible Party: Mark Wong, Westmead Medical Oncology
Other Study IDs: MWWH009
Record Dates: First submitted 2010-03-01; First posted 2010-03-02 (Estimated); Last update posted 2010-03-02 (Estimated); Status verified 2010-02

CONDITIONS: Hepatocellular Cancer
Keywords: Patients with advanced hepatocellular cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- HCC patients on Sorafenib

SUMMARY:
Sorafenib improves overall survival and progression free survival in advanced hepatocellular carcinoma. Wide interindividual pharmacokinetic variability was observed. Data from early phase trials in solid tumours showed trough sorafenib levels were associated with incidence of skin rash and hypertension. Rash, hypertension and higher trough levels were moderately predictive of progression free survival.The trough level of sorafenib may be predictive of survival and response in patients treated with sorafenib for advanced hepatocellular carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* ECOG ≤ 2
* Histologically or cytologically diagnosed hepatocellular carcinoma, or diagnosis on at least one cross-sectional imaging with the characteristic appearance of HCC (i.e. liver lesion with arterial enhancement and portal venous washout)
* Decision to treat with single agent sorafenib at 400mg bid (dose reductions or interruptions are permitted if side effects occur during treatment)
* No prior systemic chemotherapy or targeted therapy
* Child-Pugh liver function class A or B
* At least one untreated target lesion that can be measured in one dimension according to RECIST
* Adequate organ functions

Exclusion Criteria:

* Prior systemic chemotherapy or molecularly targeted therapy
* Concurrent active malignancy
* Concomitant strong CYP3A4 induced or inhibitor at a therapeutic dose (see section 6.4.1)
* Medical or psychiatric conditions that compromise the patient's ability to give informed consent
* Hypertension that cannot be controlled by medications (> 150/100 mmHg despite optimal medical therapy)
* History of, or known brain metastases (skull metastases allowed), carcinomatous meningitis, or leptomenigeal disease
* Major surgery (e.g. open abdominal therapy, pelvic, thoracic, orthopaedic or neurosurgery) within 4 weeks of the date of first dose
* Local-regional treatment (i.e. percutaneous and trans-arterial procedures) within 4 weeks. Restaging CT or MRI scan must be repeated at least 4 weeks after local-regional treatment and within 3 weeks before the date of first dose
* For patients treated with Yttrium (90Y) radiotherapy, a washout period of 2 months is required.
* Evidence of severe or uncontrolled systemic disease or any concurrent condition which in the investigator's opinion makes it undesirable for the patient to participate in the study or which would jeopardize compliance with the protocol
* Pregnancy or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with advanced HCC who are to commence Sorafenib
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2010-02; Primary Completion 2012-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
To demonstrate the correlation of trough sorafenib level with overall survival in advanced hepatocellular carcinoma | 4 years

SECONDARY OUTCOMES:
To correlate trough sorafenib level with progression free survival | 4 years
To correlate trough sorafenib level with response (disease-control vs progressive disease) by RECIST criteria | 4 years
To correlate trough sorafenib level with alpha fetoprotein (AFP) response | 4 years
To correlate trough sorafenib level with side effects (rash and hypertension) | 4 years

CONTACTS AND LOCATIONS:
Locations (1):
- Westmead Hospital, Westmead, New South Wales, Australia